CLINICAL TRIAL: NCT06807593
Title: Treatment of Immune Checkpoint Inhibitor-related Diarrhea and/ or Colitis With Ustekinumab in Cancer Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0417; NCI-2025-00795 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Participants will be identified per the evaluation of primary oncology and/or gastroenterology consult services.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — Given by infusion

SUMMARY:
The goal of this clinical research study is to learn if ustekinumab can help to control immune-related diarrhea and/or colitis in cancer patients.

DETAILED DESCRIPTION:
Primary Objectives:

To assess the efficacy of ustekinumab for clinical remission/response of immune-related diarrhea and/or colitis

To assess the efficacy of ustekinumab in reducing fecal calprotectin levels

Secondary Objectives:

To assess steroid free IMDC remission by week 4 and 8

To assess the IMDC recurrence by week 4 and 8

To assess the time duration to IMDC recurrence and overall survival

To assess the efficacy of ustekinumab to achieve endoscopic remission of immune-related diarrhea and/or colitis

To identify immune signatures related to GI irAEs and those specific to responsiveness to ustekinumab

To identify pro-inflammatory immune signatures in serum

To assess patient symptom and QOL

ELIGIBILITY:
Inclusion Criteria:

1. Patients who receive any type of ICI therapy
2. Patients with ≥ grade 2 immune-related diarrhea and/or colitis according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 within 45 days prior to enrollment in study
3. Patients with ability to understand and willingness to sign informed consent
4. Patients with a diagnosis of any type of solid tumors on ICI systemic therapy
5. No concern for active concomitant GI infection for immune-related diarrhea and/or colitis work up at the time of protocol therapy initiation as confirmed by stool tests or as per the treating physician based on clinical presentation
6. Patient who has been cleared for enrollment by Infectious Diseases consultant or treating physician if positive infection workup or screening tests (e.g. lifelong positive T- spot due to BCG inoculation, chronic colonization) prior to initiation of diarrhea/colitis treatment and/ or imaging (e.g. CXR, CT CAP etc) confirms the absence of active infections (e.g. TB) within 60 days prior to initiation of protocol therapy
7. Concurrent or prior cancer therapy (non-checkpoint inhibitors) that are not deemed as a significant contributor of the GI adverse event can be allowed in the study.
8. Patients can be on the steroid treatment within 45 days before Ustekinumab
9. Patients with non- GI immune-related adverse events (irAEs) can be enrolled if there is no contraindication to the use of ustekinumab in the treatment of the non-GI irAEs present
10. Patients with a new index event of . grade 2 immune-related diarrhea and/or colitis may be enrolled if previous IMDC event was . 1 year ago with successful treatment and clinical remission

Exclusion Criteria:

1. Patients younger than 18 years of age
2. Patients with persistent gastrointestinal infection confirmed with positive testing despite completing 5 days of antibiotics
3. Patients with history of inflammatory bowel disease and/or radiation enterocolitis with active disease status at the time of study treatment initiation
4. Pregnant and breastfeeding women
5. Women of child-bearing potential who have positive urine or serum pregnancy test or refuse to do pregnancy test unless last menstrual cycle was > 1 year prior to consent and/ or clear documentation states that patient is peri- or post-menopausal or there was recent supporting objective evidence of 'no pregnancy' status (e.g. blood or imaging) within 30 days prior to enrollment in study
6. Patients who develop concurrent non-GI toxicity (irAEs) at the time of study treatment initiation, with contraindication to the use of ustekinumab in the treatment of the non GI irAEs present
7. Patients have already received other biologic treatment for IMDC such as infliximab, vedolizumab, EXCEPT if these drugs were used in a previous IMDC event that occurred ≥ 1 year earlier at which time there was complete resolution of the disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Yinghong Wang, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org